CLINICAL TRIAL: NCT00322907
Title: A Randomised Safety and Efficacy Trial of Rifampicin/Cotrimoxazole/Isoniazid Versus Mefloquine or Quinine+SP Against Resistant Malaria in Papua New Guinea
Brief Title: Cotrifazid Safety and Efficacy Against Malaria
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Center for Primary Care and Public Health (Unisante), University of Lausanne, Switzerland (Other)
Collaborators: Papua New Guinea Institute of Medical Research (Other Government); Swiss Tropical & Public Health Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Fatol 1
Record Dates: First submitted 2006-05-05; First posted 2006-05-08 (Estimated); Last update posted 2006-05-08 (Estimated); Status verified 1999-10

CONDITIONS: Clinical Malaria
Keywords: malaria; treatment; cotrifazid; clinical trial; efficacy
MeSH Terms: conditions — Malaria

INTERVENTIONS:
Drug: Cotrifazid vs mefloquine or quinine+SP

SUMMARY:
The purpose of this study was to assess the safety and efficacy of Cotrifazid to treat uncomplicated resistant malaria and to compare the outcome with mefloquine or quinine+sulfadoxine/pyrimethamine (SP)

DETAILED DESCRIPTION:
Design: Open-label, block-randomised, comparative, multicentric trial. Setting: Four primary care health facilities, two in urban and two in rural areas of Madang and East Sepik Province, Papua New Guinea.

Participants: Patients of all ages with recurrent uncomplicated malaria Intervention: Random assignment to receive either Cotrifazid, mefloquine or the standard treatment of quinine+sulfadoxine/pyrimethamine (SP).

Outcome measures: Incidence of clinical and laboratory adverse events; rate of clinical and/or parasitological failure at day 14

ELIGIBILITY:
Inclusion Criteria:

All subjects > 6 months of age who presented at the centres and who were diagnosed with malaria (history of fever, OptiMAL® test positive, no other major symptom) and who had already been treated for malaria in the 28 days before, could be included in the study, if the subject or legal guardian (for children) gave informed consent and if the clinician in charge would have given the standard treatment for resistant malaria independent of the study -

Exclusion Criteria:

A subject was not to be included if the clinician preferred to use quinine for whatever reason, if the patient had one of the symptoms or signs of complicated or severe malaria (i.e. history of recent convulsion, any neurological sign or impairment of consciousness, heavy vomiting, haemoglobinuria, respiratory distress, bleeding, circulatory collapse, shock, jaundice, haemoglobin < 5 g/dl), had contra-indications for mefloquine (history of psychiatric disorder, epilepsy), or was pregnant.

-

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 330
Dates: Start 2000-04; Study Completion 2003-01

PRIMARY OUTCOMES:
Clinical treatment failure rate on day 14.
Incidence of adverse events.

SECONDARY OUTCOMES:
Parasitological failure rate on day 14
Fever clearance time
Parasite clearance time
Symptoms clearance time
Occurrence of complications

CONTACTS AND LOCATIONS:
Overall Officials: Blaise Genton, MD, PhD, Principal Investigator — Swiss Tropical & Public Health Institute
Locations (1):
- Health centers, Madang and Maprik, Madang and East Sepik Province, Papua New Guinea